CLINICAL TRIAL: NCT06836856
Title: Evaluating the Impact of Adjuvant Use of Beta Blockers on Clinical Outcomes in Patients With Traumatic Brain Injury
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha Mansour, Associate Profesor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-37
Record Dates: First submitted 2025-01-20; First posted 2025-02-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-01

CONDITIONS: TBI Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Propranolol; Carvedilol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Arm (Placebo Comparator)
  Interventions: Drug: control
- propranolol (Active Comparator): propranolol
  Interventions: Drug: propranolol
- carvedilol (Active Comparator): Carvid (carvedilol)
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: control — Patients will receive standard care with no interventions until end of treatment.
  Arms: Control Arm
Drug: propranolol — starting at 20mg propranolol three times daily by mouth or per feeding tube. The dose was increased daily in 20mg three times daily increments (60mg/day total) until heart rate (HR) was less than 100 beats per minute (bpm) with maximum dose of 640mg/day in addition to standard care until end of treatment.
  Arms: propranolol
Drug: Carvedilol — starting at 6.25mg carvedilol three times daily by mouth or per feeding tube. The dose was increased daily in 6.25 mg three times daily increments (18.75 mg/day total) until heart rate (HR) was less than 100 beats per minute (bpm) with maximum dose of 100 mg/day in addition to standard care until end of treatment.
  Arms: carvedilol

SUMMARY:
Propranolol primarily acts as a non-selective beta blocker, blocking both beta-1 and beta-2 adrenergic receptors, while carvedilol exhibits a broader spectrum of action by also blocking alpha-1 adrenergic receptors. The receptor blockade profile of a beta blocker can influence its physiological effects and potential therapeutic benefits in TBI. Therefore, the variation in receptor selectivity may result in differences in their impact on secondary brain injury processes and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with moderate & severe TBI detected on admission by CT scan and GCS score of ≤ 13 who either do not have any other injuries or only have associated minor injuries.

Minor injuries are defined as presence of any of the following:

1. Mild intraperitoneal free fluid (IPFF) observed through abdominal ultrasound.
2. mild lung contusion detected in the chest CT scan.
3. hemothorax or pneumothorax present without accompanying symptoms of hypoxia, tachypnea, or respiratory distress.
4. simple limb fractures.

Exclusion Criteria:

1. Patients on pre-injury beta-blocker therapy.
2. Patients with any bronchospastic conditions.
3. Patients with active acute coronary syndrome.
4. TBI with GCS ≤ 13 with associated major injuries defined as the presence of any of the following:

   1. Moderate & marked IPFF requiring surgical intervention ( laparotomy ).
   2. moderate & marked lung contusion, pneumothorax & hemothorax with accompanying symptoms of hypoxia, tachypnea, lower limbs, or limb amputation.
   3. Compound fracture in the upper or lower limb.
   4. Open Faciomaxillary trauma.
5. Patients with persistent shock (systemic blood pressure <100 mmHg, base deficit > 4, or oliguria , HR < 60 b/min ) after > one week of admission.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of In-hospital mortality | 14 days
  Difference between the study grous in terms of the percentage of all-cause mortality at the end of treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Zagazig University Hospitals, Zagazig,, Zagazig
  - Zagazig University Hospitals, Zagazig

IPD SHARING:
Plan to Share IPD: No